CLINICAL TRIAL: NCT07123077
Title: Effect of Functional Exercises With Music on Older Adults With Mild Dementia
Brief Title: Functional Exercises With Music in Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Çağla ÖZGÖREN, Principal Investigator, Lecturer in Physiotherapy, Specialist Physiotherapist, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedipolU-FTR-ÇÖ-02
Record Dates: First submitted 2025-07-28; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mild Dementia; Music Therapy
Keywords: Mild Dementia; Functional Exercise; Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person who performed the statistical analysis was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Exercise Group (Experimental): The exercise program consisted of warm-up, strength-balance, and cool-down exercises, all of which were administered to the participants under the supervision of a physiotherapist. Necessary precautions were taken to prevent participants from falling during the standing balance exercises.
  Interventions: Other: Functional Exercises
- Functional Exercises with Music Group (Experimental): The exercise program was implemented with the same content, duration, and by the same researcher as the protocol used in the functional exercise group. Exercise sessions were conducted with music, and the music was provided by a single expert researcher. Slow-paced pieces in the Rast mode were selected for warm-up and cool-down exercises, while more upbeat pieces in the Mahur mode were used for strength and balance exercises. To enhance participants' concentration, instrumental compositions in these selected Turkish classical music modes were used during the sessions. Traditional Turkish instruments such as qanun, ney, kudüm, and oud were chosen to perform the compositions.
  The music pieces were recorded in a quiet environment and played for the participants during exercise sessions via a JBL Go Essential Bluetooth speaker (IPX7). The use of pre-recorded music provided a standardized auditory stimulus for all participants, increasing the reproducibility of of the intervention and cont
  Interventions: Other: Functional Exercises; Other: Music Intervention

INTERVENTIONS:
Other: Functional Exercises — Warm-Up Exercises (10 min): Diaphragmatic breathing exercise, neck rotation (right & left), rotational shoulder movements, trunk rotation, triceps stretching exercise, hamstring stretching exercise Each exercise was performed for 8 repetitions.
  Strengthening Exercises (40 min):
  In a seated position:
  Ankle plantar flexion and dorsiflexion exercises, ankle circumduction, knee extension, hip flexion, shoulder joint range of motion exercises in all directions, elbow and hand flexion-extension exercises
  In a standing position:
  Hip extension, toe raises, mini squats, standing on one leg, 360-degree turning, tandem walking exercises Each exercise was performed for 8 repetitions.
  Cool-Down Exercises (10 min): Diaphragmatic breathing exercise, neck rotation (right & left), rotational shoulder movements, trunk rotation, triceps stretching exercise, hamstring stretching exercise Each exercise was performed for 8 repetitions.
Other: Music Intervention — Slow-paced pieces in the Rast mode were selected for the warm-up and cool-down exercises, while more upbeat pieces in the Mahur mode were chosen for strength and balance exercises and played to the participants throughout the sessions alongside the exercises. To enhance participants' concentration, instrumental compositions in these selected Turkish classical music modes were used. Traditional Turkish instruments such as qanun, ney, kudüm, and oud were preferred in the performance of the compositions.
  Arms: Functional Exercises with Music Group

SUMMARY:
This study aims to explore how a functional exercise program, with or without music, affects physical function and quality of life in older adults with mild dementia. Participants were divided into two groups: one group performed functional exercises alone, while the other group performed the same exercises accompanied by music. The program was conducted twice a week for 8 weeks, with each session lasting 60 minutes. Researchers evaluated changes in balance, mobility, risk and fear of falling, hand grip strength, daily living activities, and overall quality of life before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for participants were: voluntary participation, Mini-Mental State Examination (MMSE) scores between 17 and 24 indicating mild dementia
* Residing in a nursing home, being over 65 years of age,
* Having no problems understanding verbal commands.

Exclusion Criteria:

* Diagnosis of severe and untreated hearing impairment that would prevent them from listening to music
* A history of musculoskeletal injury or neurological deficit that could affect exercise performance
* A psychiatric disorder that could interfere with exercise compliance
* Inability to cooperate during tests and exercises, and failure to attend two consecutive sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Four-Stage Balance Test | From enrollment to the end of treatment at 8 weeks
  The Four-Stage Balance Test is a static balance assessment that measures an individual's ability to maintain stability in various standing positions. In the first stage, the feet are placed side by side. In the second stage, the instep of one foot is placed next to the big toe of the other foot. The third stage involves the tandem stance, where one foot is positioned directly in front of the other, with the heel touching the toes. In the final stage, the individual is asked to stand on one foot.
  At each stage, the participant is expected to maintain the position without moving or losing stability for 10 seconds. If the feet shift or the individual requires external support, the test is terminated. Participants are allowed to progress to the next stage only if they successfully complete the current one. The highest stage successfully completed is recorded.
  The test is not administered to individuals who are at high risk of falling or cannot be safely supported.
Katz Index of Independence in Activities of Daily Living | From enrollment to the end of treatment at 8 weeks
  It measures an individual's capacity to perform activities that are commonly required in daily life and their level of dependence on others. The index evaluates six basic activities: bathing, dressing, toileting, continence, and feeding. As the total score increases, the individual's ability to carry out these functions independently also increases.

SECONDARY OUTCOMES:
Hand Grip Strength | From enrollment to the end of treatment at 8 weeks
  To assess the maximum isometric contraction strength of the hand and forearm muscles, a Camry digital hand dynamometer (Model EH101, Zhongshan Camry Electronic Co., Ltd., Zhongshan, China) was used. The measurement was conducted in accordance with the protocol recommended by the American Society of Hand Therapists for standardized hand grip strength assessment. Participants were seated in a comfortable position with their feet shoulder-width apart. Shoulders were in neutral rotation and vertical adduction. The dominant elbow was flexed at 90°, forearms were in a neutral position, and the wrist was positioned at 0°-30° extension and 0°-15° ulnar deviation. After achieving proper posture, participants were instructed to perform a maximal grip for 5 seconds. The measurement was repeated three times, and the average value was recorded.
World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD) | From enrollment to the end of treatment at 8 weeks
  Participants' quality of life was assessed using the World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD). The scale consists of 24 Likert-type items grouped into six subscales: sensory abilities, autonomy, past, present and future activities, social participation, death and dying, and intimacy. Higher scores on the scale indicate better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çelik, Principal Investigator — Istanbul Huzur Hospital and Dinlenme Evleri Foundation and Atlas Nursing Home; Çağla Özgören, Principal Investigator — Medipol University; Sena Özdemir Görgü, Principal Investigator — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Atlas Nursing Home, Istanbul
  - Istanbul Huzur Hospital ve Dinleme Evleri Foundation, Istanbul

IPD SHARING:
Plan to Share IPD: No